CLINICAL TRIAL: NCT07062133
Title: Clinical Evaluation of Electrical Pudendal Nerve Stimulation in Children With Postoperative Neurogenic Lower Urinary Tract Dysfunction Secondary to Tethered Cord Syndrome
Brief Title: Effectiveness of Electrical Pudendal Nerve Stimulation for Neurogenic Lower Urinary Tract Dysfunction in Pediatric Tethered Cord Syndrome Post-Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Collaborators: Shanghai Pudong Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: pdzyy-2025-07
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Neurogenic Lower Urinary Tract Dysfunction Secondary to Tethered Cord Syndrome
Keywords: Neurogenic Lower Urinary Tract Dysfunction; Tethered Cord Syndrome; Electrical Pudendal Nerve Stimulation
MeSH Terms: conditions — Neural Tube Defects

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Conventional conservative treatment including medications (e.g., oxybutynin), clean intermittent catheterization, and diaper use as needed, without EPNS intervention.
  Interventions: Other: Conventional conservative treatment
- EPNS group (Experimental): Electrical Pudendal Nerve Stimulation (EPNS) delivered by four deep acupuncture needles targeting bilateral sacrococcygeal points near the pudendal nerve. Connected to G6805-2 electrical stimulator, 2 Hz, 60 minutes/session, three times per week for 4 weeks.
  Apart from EPNS, intervention administered in this group also include conventional conservative treatment as sama as in the control group
  Interventions: Procedure: Electrical pudendal nerve stimulation; Other: Conventional conservative treatment

INTERVENTIONS:
Procedure: Electrical pudendal nerve stimulation — Electrical Pudendal Nerve Stimulation (EPNS) delivered by four deep acupuncture needles targeting bilateral sacrococcygeal points near the pudendal nerve. Connected to G6805-2 electrical stimulator, 2 Hz, 60 minutes/session, three times per week for 4 weeks.
  Arms: EPNS group
Other: Conventional conservative treatment — Conventional conservative treatment including medications (e.g., oxybutynin), clean intermittent catheterization, and diaper use as needed

SUMMARY:
The goal of this prospective observational study is to evaluate whether the addition of electrical pudendal nerve stimulation (EPNS) to standard conservative treatment can improve bladder function in pediatric patients with postoperative neurogenic bladder secondary to tethered cord syndrome . The study population consists of 50 children diagnosed with neurogenic bladder of various etiologies.

The main questions this study aims to answer are:

Does EPNS lead to significant improvement in neurogenic bladder symptom scores?

How does EPNS affect secondary clinical outcomes such as renal function, post-void residual volume, urinary leakage, and vesicoureteral reflux?

Researchers will compare clinical indicators before and after the addition of EPNS, on the background of consistent conservative management, to assess its therapeutic contribution.

Participants will:

Receive routine conservative therapy for neurogenic bladder (e.g., medications, bladder training)

Undergo EPNS sessions over a specified treatment period

Be evaluated using standardized scales and imaging or laboratory tests to monitor changes in bladder and renal function

The study will also explore whether treatment effects differ by underlying cause or symptom pattern.

DETAILED DESCRIPTION:
This prospective, controlled clinical study aims to evaluate the therapeutic efficacy of "sacral four-needle" electrical pudendal nerve stimulation (EPNS) in children with neurogenic lower urinary tract dysfunction (NLUTD) following surgical untethering for tethered cord syndrome (TCS). TCS is a common spinal dysraphism in pediatrics, often resulting in bladder dysfunction postoperatively despite timely surgical intervention. Conventional management, including intermittent catheterization and pharmacotherapy, carries limitations such as poor adherence and persistent symptoms. EPNS, a non-invasive acupuncture-based neuromodulation technique targeting the pudendal nerve via anatomically guided deep needling and low-frequency electrical stimulation, has shown promise in adult neurogenic bladder cases. This study will enroll approximately 50 children aged 3-18 with confirmed TCS and persistent NLUTD after initial surgery. Participants will be assigned to receive either routine conservative therapy alone or combined with EPNS over a four-week period (three sessions per week). Treatment efficacy will be assessed through changes in the Neurogenic Bladder Symptom Score (NBSS), along with secondary endpoints including post-void residual volume, voiding frequency, episodes of incontinence, renal function, and incidence of urinary tract infections. Follow-up will continue for six months post-treatment to evaluate sustained effects. The study employs blinded outcome assessment, with standardized protocols for needling, stimulation parameters, and symptom tracking. It further includes subgroup analyses based on disease etiology and symptom type (storage vs. voiding dysfunction). The research integrates traditional acupuncture with neuroanatomical precision and modern bladder rehabilitation theory, aiming to establish a replicable, low-cost, and scalable pediatric bladder dysfunction intervention model. By addressing a current gap in pediatric urological rehabilitation, the study seeks to contribute evidence toward standardizing EPNS as a viable adjunct therapy in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-18 years
* Diagnosed with TCS (by spinal MRI) and NLUTD (by urodynamic study)
* First-time detethering surgery completed
* Be able to comply with acupuncture treatment and follow-up
* Informed consent obtained from legal guardian

Exclusion Criteria:

* Severe systemic diseases
* Current urinary tract infection, severe VUR, hydronephrosis, structural obstruction
* Prior aggressive urological surgery (e.g., augmentation cystoplasty)
* Prior or planned pudendal/sacral nerve implant
* Botulinum toxin injection within past 12 months
* Planned reoperation within 6 months

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Neurogenic Bladder Symptom Score (NBSS) from baseline to 4 weeks post-treatment | Baseline to 4 weeks (end of treatment)
  The Neurogenic Bladder Symptom Score (NBSS) is a validated, patient-reported questionnaire specifically designed to evaluate urinary symptoms and quality of life in individuals with neurogenic lower urinary tract dysfunction (NLUTD). It includes domains assessing incontinence, storage and voiding symptoms, complications (such as infections or catheter use), and the impact on daily life. In this study, the NBSS will be administered at baseline (prior to treatment initiation) and again after the 4-week intervention period. The primary outcome measure will be the change in total NBSS score between these two time points. A decrease in NBSS score reflects symptom improvement. Assessments will be completed by participants or their guardians under guidance from trained study personnel.

SECONDARY OUTCOMES:
Serum creatinine and estimated glomerular filtration rate (eGFR) | Baseline, 4 weeks, and 6-month follow-up
  Serum creatinine and estimated glomerular filtration rate (eGFR) are standard laboratory measures used to evaluate renal function. Serum creatinine reflects the concentration of creatinine in the blood, a waste product filtered by the kidneys, while eGFR provides an estimate of kidney filtration efficiency adjusted for age, sex, and body size.
Change in post-void residual urine volume (PVR) | Baseline, after 5th session, 10th session, end of treatment (week 4), and at 2-, 4-, 6-month follow-up
  Post-void residual urine volume (PVR) is a clinical parameter used to assess the efficiency of bladder emptying. It is defined as the amount of urine remaining in the bladder immediately after voluntary urination. In this study, PVR will be measured using noninvasive bladder ultrasound (portable or bedside ultrasound device) performed by trained personnel.A reduction in PVR indicates improved bladder emptying function, which is a critical component of managing NLUTD.
Urinary leakage volume | Baseline to 4 weeks, and at 2-, 4-, and 6-month follow-up
Incidence or grade of vesicoureteral reflux (VUR) | Baseline and 6-month follow-up
  Vesicoureteral reflux (VUR) is the retrograde flow of urine from the bladder into the ureters and potentially the kidneys, which can contribute to recurrent urinary tract infections and renal damage.The outcome will include (1) the presence or absence of VUR and (2) any change in VUR grade among participants with reflux at baseline. The primary interest is in identifying any improvement (reduction in grade or resolution) or worsening of VUR following the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pudong Hospital of Traditional Chinese Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
This is an early-phase, single-center exploratory trial with a limited sample size. The primary goal is to generate pilot data for future large-scale studies. At present, there is no confirmed plan to share de-identified individual participant data (IPD). However, data sharing may be considered in the future depending on study outcomes, ethical approvals, and publication status.
  If data are made available in the future, access will be provided to qualified researchers upon reasonable request and subject to institutional data use agreements and ethical oversight.